CLINICAL TRIAL: NCT06902545
Title: Post-marketing Observational Study of VYLOY (Zolbetuximab) Injection 100 mg for Locally Advanced Unresectable or Metastatic Gastric or Gastroesophageal Junction (GEJ) Adenocarcinoma in South Korea
Brief Title: A Study to Observe the Safety of VYLOY (Zolbetuximab) in People in South Korea With Gastric or Gastroesophageal Junction Cancer.
Status: Recruiting | Type: Observational
Sponsor: Astellas Pharma Korea, Inc. (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Other Study IDs: 8951-PV-0001
Record Dates: First submitted 2025-03-24; First posted 2025-03-30 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Locally Advanced Unresectable Gastroesophageal Junction (GEJ) Adenocarcinoma or Cancer; Locally Advanced Unresectable Gastric Adenocarcinoma or Cancer; Metastatic Gastric Adenocarcinoma or Cancer; Metastatic Gastroesophageal Junction (GEJ) Adenocarcinoma
Keywords: Locally Advanced Unresectable Gastroesophageal Junction (GEJ) Adenocarcinoma Cancer; Locally Advanced Unresectable Gastric Adenocarcinoma Cancer; Metastatic Gastric Adenocarcinoma Cancer; Metastatic Gastroesophageal Junction (GEJ) Adenocarcinoma; Claudin 18.2; Human epidermal growth factor receptor 2 (HER2) Negative; zolbetuximab; Pharmcovigilence
MeSH Terms: conditions — Adenocarcinoma; Neoplasms | interventions — zolbetuximab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Vyloy: Patients who receive treatment with Vyloy injection 100 mg (zolbetuximab), according to the approved local label.
  Interventions: Drug: zolbetuximab

INTERVENTIONS:
Drug: zolbetuximab — Intravenous
  Other Names: Vyloy

SUMMARY:
This study is for people in South Korea who have cancer in or around the stomach (gastric cancer) or cancer where the food pipe (esophagus) joins the stomach, called gastroesophageal junction (GEJ) cancer. Their cancer is locally advanced, unresectable, or metastatic. Locally advanced means the cancer has spread to tissue close by. Unresectable means the cancer cannot be removed by surgery. Metastatic means the cancer has spread to other parts of the body.

In South Korea, VYLOY is approved for the treatment of gastric cancer or GEJ cancer. The people in this study will receive VYLOY as part of their usual treatment for their cancer. In standard clinical practice VYLOY is given to people slowly through a tube into a vein.

The main aim of the study is to collect information in a real-world setting about the safety of VYLOY in people with gastric cancer or GEJ cancer in clinics in South Korea. This study will also help researchers learn how long people's gastric cancer or GEJ cancer stays stable.

This study is about collecting information only. This is known as an observational study. The individual's doctor decides on treatment, not the sponsor (Astellas). The study will last about 1 year (54 weeks).

ELIGIBILITY:
Inclusion Criteria:

* Patients who receive treatment with VYLOY injection, according to the approved local label.

Exclusion Criteria:

* Patients with any contraindication for VYLOY injection, according to the approved local label.
* Patients who are registered or scheduled to be registered in any clinical trials involving investigational drug administration.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who have locally advanced unresectable or metastatic HER2-negative, and CLDN18.2-positive, gastric or GEJ adenocarcinoma who are prescribed VYLOY injection in combination with fluoropyrimidine- and platinum-containing chemotherapy for the first line treatment in South Korea.
Sampling Method: Non-Probability Sample
Enrollment: 377 (Estimated)
Dates: Start 2025-04-03 (Actual); Primary Completion 2030-07-31 (Estimated); Study Completion 2030-07-31 (Estimated)

PRIMARY OUTCOMES:
Number of patients with an adverse event (AE) | Up to 54 Weeks after the first administration of VYLOY
  Adverse events (AEs) will be coded using MedDRA. An AE is defined as any untoward medical occurrence in a patient administered a study drug, and which does not necessarily have to have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a medicinal product whether or not considered related to the medicinal product.
Number of patients with an adverse drug reaction (ADR) | Up to 54 Weeks after the first administration of VYLOY
  An ADR is defined as any noxious and unintended response associated with the use of a drug in humans, at any dose, where a causal relationship is at least a reasonable possibility.
Number of patients with a serious AE (SAE) | Up to 54 Weeks after the first administration of VYLOY
  An AE is considered "serious" if, in the view of either the investigator or sponsor, the event: results in death, is life-threatening, requires hospitalization or prolongation to hospitalization results in persistent or significant disability or incapacity, results in congenital anomaly or birth defect, or other medically important event.
Number of patients with a serious ADR (SADR) | Up to 54 Weeks after the first administration of VYLOY
  An ADR considered "serious" if, in the view of either the investigator or sponsor, the event: results in death, is life-threatening, requires hospitalization or prolongation to hospitalization results in persistent or significant disability or incapacity, results in congenital anomaly or birth defect, or other medically important event.
Number of patients with an unexpected AE (UAE) | Up to 54 Weeks after the first administration of VYLOY
  An UAE is an AE that the nature or severity of which is not consistent with the information in the Precautions in Use Section of approved Korean label.
Number of patients with an unexpected ADR (UADR) | Up to 54 Weeks after the first administration of VYLOY
  An UADR is defined as an unexpected adverse drug reaction.
Number of patients who died during the study | Up to 54 Weeks after the first administration of VYLOY
Number patients with an AE leading to death | Up to 54 Weeks after the first administration of VYLOY
Number of patients with an important risk compared to number of patients evaluated | Up to 54 Weeks after the first administration of VYLOY
  An important risk is classified as an important identified risk and an important potential risk.
  An identified risk is defined as the risk that correspond to undesirable clinical outcomes, with sufficient scientific evidence that the undesirable clinical outcome is caused by the drug. "Important Identified Risks" are identified risks that have the potential to affect the risk-benefit balance of a product.
  An potential risk is defined as the risk that correspond to undesirable clinical outcomes, with some, but not sufficient, evidence to estimate that the undesirable clinical outcome is caused by the drug. "Important Potential Risks" are potential risks that have the potential to affect the risk-benefit balance of a product.

SECONDARY OUTCOMES:
Progression free survival (PFS) | Up to 54 Weeks after the first administration of VYLOY
  PFS is defined as time from start of VYLOY to progressive disease (PD) or death from any cause, whichever occurs first.

CONTACTS AND LOCATIONS:
Overall Officials: Central Contact, Study Director — Astellas Pharma Korea, Inc.
Locations (12):
- South Korea (12):
  - KR82010, Goyang-si, Gyeonggi-do
  - KR82008, Suwon, Gyeonggi-do
  - KR82006, Yangsan, Gyeongsangnam-do
  - KR82012, Hwasun Gun, Jeollanam-do
  - KR82001, Seoul
  - KR82002, Seoul
  - KR82003, Seoul
  - KR82004, Seoul
  - KR82005, Seoul
  - KR82007, Seoul
  - KR82011, Seoul
  - KR82013, Seoul

IPD SHARING:
Plan to Share IPD: No
Access to anonymized individual participant level data will not be provided for this trial. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.